CLINICAL TRIAL: NCT00065884
Title: Valproate Response in Aggressive Autistic Adolescents
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: P30HD002528 (NIH); K08MH001516 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-06

CONDITIONS: Autism
Keywords: Adolescents
MeSH Terms: conditions — Autistic Disorder | interventions — Valproic Acid

INTERVENTIONS:
Drug: Valproate

SUMMARY:
This study will examine the effect of valproate, a medication used to treat seizures and bipolar disorder, on aggressive behavior in children and adolescents with autism.

DETAILED DESCRIPTION:
Autism is a complex biological disorder that generally lasts throughout a person's life. It starts before age three and causes delays or problems with many different ways in which a person develops or grows. Some people with autism become very aggressive and can hurt others or themselves. This study will test the hypothesis that aggressive autistic adolescents will show a significantly greater response to valproate maintained at blood levels of 75-100 mcg/ml than to placebo. The study will also assess the safety of valproate in autistic adolescents. This represents the first double-blind study of valproate in mentally retarded/developmentally delayed populations.

Participants in this study will undergo DSM-IV evaluation, the Autism Diagnostic Interview-Revised and Autism Diagnostic Observation Schedule, and baseline blood tests. After baseline screening, all participants will be given a placebo for 1 week. Participants will then be randomized to receive either valproate or placebo for 8 weeks. Dosage adjustment according to blood levels drawn at the end of weeks 2 and 4 will be arranged with parents by a child psychiatrist without breaking the blind. The Aberrant Behavior Check-list-Community (ABC-C) irritability subscale will be the primary measure; the Overt Aggression Scale (OAS), ABC-C hyperactivity subscale, Clinical Global Impressions (CGI) problem severity, Self-Injurious Behavior Questionnaire (SIB-Q), and a valproate side effects checklist will be secondary measures.

ELIGIBILITY:
Inclusion Criteria

* Autism
* Lives in the Kansas City area

Exclusion Criteria

* Psychoactive maintenance medication
* Degenerative central nervous system disorder
* Unstable medical illness
* Seizures in the 6 months prior to study entry
* History of valproate sensitivity or previous liver disease
* History of ovarian cysts
* Low platelet count or raised liver transaminases

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30

CONTACTS AND LOCATIONS:
Overall Officials: Jessica A. Hellings, M.D., Principal Investigator — University of Kansas
Locations (1):
- Outpatient MR/Autism Clinic, University of Kansas, Kansas City, Kansas, United States